CLINICAL TRIAL: NCT00045032
Title: A Randomized Three-Arm, Multicenter Comparison of 1 Year and 2 Years of Herceptin Versus No Herceptin in Women With HER2-Positive Primary Breast Cancer Who Have Completed Adjuvant Chemotherapy
Brief Title: Herceptin (Trastuzumab) in Treating Women With Human Epidermal Growth Factor Receptor (HER) 2-Positive Primary Breast Cancer
Acronym: HERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Breast International Group (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); NCIC Clinical Trials Group (Network); ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO16348; BIG-01-01; EU-20216; ROCHE-B016348E; ROCHE-B016348C; EORTC-10011; CAN-NCIC-MA24; IBCSG-28-02
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (3):
- Observation Arm (No Intervention): Participants who have completed definitive surgery and systemic adjuvant chemotherapy will be observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant. No Herceptin will be provided.
- Herceptin 1-Year Arm (Experimental): Participants who have completed definitive surgery and systemic adjuvant chemotherapy will receive Herceptin for 1 year or until disease recurrence, whichever occurs first. Participants will be observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant.
  Interventions: Drug: Herceptin
- Herceptin 2-Year Arm (Experimental): Participants who have completed definitive surgery and systemic adjuvant chemotherapy will receive Herceptin for 2 years or until disease recurrence, whichever occurs first. Participants will be observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — Herceptin will be given as a loading dose of 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion on Day 1, followed by a maintenance dose of 6 mg/kg via IV infusion 3 weeks later and thereafter every 3 weeks.
  Other Names: Trastuzumab
  Arms: Herceptin 1-Year Arm
Drug: Herceptin — Herceptin will be given as a loading dose of 8 mg/kg via IV infusion on Day 1, followed by a maintenance dose of 6 mg/kg via IV infusion 3 weeks later and thereafter every 3 weeks.
  Other Names: Trastuzumab
  Arms: Herceptin 2-Year Arm

SUMMARY:
The purpose of this trial is to evaluate Herceptin treatment for 1 year and 2 years (versus observation/no Herceptin) in women with HER2-overexpressing primary breast cancer who have completed (neo-)adjuvant systemic chemotherapy, definitive surgery, and radiotherapy, if applicable. Efficacy and safety will be assessed for 10 years from randomization for each participant. All participants will continue to be followed for survival until 10 years after enrollment of the last participant.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic primary invasive breast cancer overexpressing HER2 (determined by immunohistochemistry 3+ or positive fluorescence in situ hybridization test) that has been histologically confirmed, adequately excised, axillary node positive or negative, and tumor size at least T1c according to Tumor/Node/Metastasis (TNM) staging
* Completion of at least 4 cycles of (neo-)adjuvant systemic chemotherapy, definitive surgery, and radiotherapy, if applicable
* Known hormone receptor status
* Baseline left ventricular ejection fraction (LVEF) greater than or equal to (≥) 55 percent (%)

Exclusion Criteria:

* Prior invasive breast carcinoma
* Other malignancies except for curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Clinical T4 tumors
* Cumulative doxorubicin exposure greater than (>) 360 milligrams per meter-squared (mg/m^2) or epirubicin >720 mg/m^2 or any prior anthracyclines unrelated to the present breast cancer
* Peripheral stem cell or bone marrow stem cell support
* Prior mediastinal irradiation except for internal mammary node irradiation for the present breast cancer
* Non-irradiated internal mammary nodes or supraclavicular lymph node involvement
* Prior anti-HER2 therapy for any other reason or other prior biologic or immunotherapy for breast cancer
* Concurrent anti-cancer treatment in another investigational trial
* Serious cardiac or pulmonary conditions/illness, or any other conditions that could interfere with planned treatment
* Poor hematologic, hepatic, or renal function
* Pregnancy or lactation
* Women of childbearing potential or less than 1 year post-menopause unwilling to use adequate contraceptive measures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5099 (Actual)
Dates: Start 2001-11; Primary Completion 2005-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martine J. Piccart-Gebhart, MD, PhD, Study Chair — Jules Bordet Institute; Robert E. Coleman, MD, FRCP, Study Chair — Cancer Research Centre at Weston Park Hospital; Karen A. Gelmon, MD, Study Chair — British Columbia Cancer Agency; Kathleen I. Pritchard, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Olivia Pagani, MD, Study Chair — Ospedale Beata Vergine
Locations (203):
- Hospital Aleman de Buenos Aires, Buenos Aires, Buenos Aires, Argentina
- Australia (4):
  - Saint John of God Hospital, Geelong, Australian Capital Territory
  - Toowoomba Hospital, Toowoomba, Queensland
  - Andrew Love Cancer Centre, Geelong, Victoria
  - Mount Hospital, Perth, Western Australia
- Austria (11):
  - Landeskrankenhaus Feldkirch, Feldkirch-Tisis
  - Innsbruck Universitaetsklinik, Innsbruck
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - St. Vincent's Hospital, Linz Donau
  - Landeskrankenanstalten - Salzburg, Salzburg
  - Landeskrankenhaus St. Poelten, Sankt Pölten
  - Universitaetsklinik fuer Innere Medizin I, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
  - LKH Villach, Villach
  - LKH Voecklabruck, Vöcklabruck
  - A. oe. Krankenhaus Wiener Neustadt, Wiener Neustadt
- Belgium (14):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Reseau Hospitalier De Medecine Sociale, Baudour
  - Hopital Universitaire Erasme, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Notre Dame - Reine Fabiola, Charleroi
  - Cazk Groeninghe - Campus St-Niklaas, Kortrijk
  - Centre Hospitalier Universitaire de Tivoli, La Louvière
  - U.Z. Gasthuisberg, Leuven
  - Clinique Saint-Joseph, Liège
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Clinique Sainte Elisabeth, Namur
  - Hospital Serruys Ziekenhuis, Ostend
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Brazil (5):
  - Porto Alegre Hospital, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital Santa Rita, Porto Alegre
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Faculdade De Medicina Do ABC, Santo André
- Canada (19):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Royal Victoria Hospital of Barrie, Barrie, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Trillium Health Centre - Mississauga Site, Mississauga, Ontario
  - Algoma Regional Cancer Program at Sault Area Hospital, Sault Ste. Marie, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Prince Edward Island Cancer Centre at Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Chile (5):
  - Fundacion Arturo Lopez Perez, Santiago
  - Hospital Clinico San Borja Arriaran, Santiago
  - Hospital Dr. Sotero Del Rio, Santiago
  - Hospital Militar, Santiago
  - Instituto Nacional Del Cancer, Santiago
- China (3):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Tongji Medical University, Wuhan
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- Clinical Hospital Center Split, Split, Croatia
- Denmark (5):
  - Centralsygehus I Esbjerg, Esbjerg
  - Herning Central Hospital, Herning
  - Hillerod Hospital, Hillerød
  - Centralsygehuset I Naestved, Næstved
  - Sonderborg Sygehus, Sønderborg
- France (3):
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Clinique Claude Bernard, Metz
- Germany (15):
  - Charite - Campus Charite Mitte, Berlin
  - Evangelisches Bethesda Krankenhaus GmbH, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Martin Luther Universitaet, Halle
  - Henriettenstiftung Krankenhaus, Hanover
  - Universitaets-Hautklinik Heidelberg, Heidelberg
  - St. Vincentius-Kliniken, Karlsruhe
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Kreiskrankenhaus Leonberg - Frauenklinik, Leonberg
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Frauenklinik Vom Roten Kreuz, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Frauenklinik - Universitaetsklinikum Rostock am Klinikum Sudstadt, Rostock
  - Universitaet Ulm, Ulm
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
- Greece (2):
  - University of Crete School of Medicine, Heraklion, Crete
  - Evaggelismos Hospital, Athens
- Guatemala (2):
  - Centro Medico, Guatemala City
  - Hospital Roosevelt, Guatemala City
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Hungary (3):
  - Semmelweis University, Budapest
  - National Institute of Oncology, Budapest
  - Fovarosi Onkormanyzat Szent Margit Korhaz, Okologia, Budapest
- Cork University Hospital, Cork, Ireland
- Sieff Hospital, Safed, Israel
- Italy (32):
  - Ospedale San Lazzaro, Alba
  - Ospedale Presenti Fenaroli, Alzano Lombardo
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale degli Infermi - ASL 12, Biella
  - Ospedale Bellaria, Bologna
  - Spedali Civili di Brescia, Brescia
  - Ospedale Oncologico A. Businco, Cagliari
  - Ospedale B. Ramazzini, Carpi
  - Ospedale Valduce, Como
  - Ospedale Santa Croce, Cuneo
  - Universita Degli Studi Di Florence, Firenze (Florence)
  - Azienda Ospedaliero Careggi, Florence
  - Morgagni-Pierantoni Ospedale, Forlì
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospedale A. Manzoni, Lecco
  - Presidio Ospedaliero, Livorno
  - Carlo Poma Hospital, Mantova
  - European Institute of Oncology, Milan
  - Ospedale Niguarda Ca'Granda, Milan
  - University of Modena Hospital and Reggio Emilia School of Medicine, Modena
  - Azienda Ospedaliera Di Parma, Parma
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - Policlinico Monteluce, Perugia
  - Azienda Ospedaliera, Reggio Emilia
  - Ospedale San Filippo Neri, Rome
  - Ospedale Sant' Eugenio, Rome
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale Civile ASL 1, Sassari
  - Primario U.O. di Oncologia Medica, Trento
  - Ospedale Ostetrico Ginecologica Sant Anna, Turin
  - Universita di Torino, Turin
- Japan (2):
  - Tokai University School Of Medicine, Kanagawa
  - Tokyo Metropolitan - Komagome Hospital, Tokyo
- Netherlands (3):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Maasland Hospital, Sittard
  - Diakonessenhuis Utrecht, Utrecht
- Poland (4):
  - Medical University of Gdansk, Gdansk
  - Oncologic Center, Gliwice
  - Medical University, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (6):
  - Instituto Portugues de Oncologia, Centro Regional de Coimbra, Coimbra
  - Hospitais da Universidade de Coimbra (HUC), Coimbra
  - Maternidade Byssaia Barreto, Coimbra
  - Hospital Distrital De Faro, Faro
  - Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon
  - University Hospital of Santa Maria, Lisbon
- Russia (2):
  - Moscow Oncology Hospital, Moscow
  - P.A. Hertzen Research Oncology Institute, Moscow
- Johns Hopkins Singapore International Medical Centre, Singapore, Singapore
- South Africa (5):
  - Groote Schuur Hospital, Cape Town
  - Parklands Hospital, Durban
  - Sandton Oncology Centre, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Pretoria - East Hospital, Lynnwood
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center at Yonsei University Medical Center, Seoul
- Spain (20):
  - Centro Oncologico De Galicia Jose Antonio Quirogay Pineyro, A Coruña
  - Hospital De La Ribera, Alzira
  - Hospital Del Mar, Barcelona
  - Hospital Universitario San Cecilio de Granada, Granada
  - Hospital General Universitario De Guadalajara, Guadalajara
  - Hospital Juan Ramon Jimenez, Huelva
  - Hospital Cuidad de Jaen, Jaén
  - Hospital Insular de Gran Canaria, Las Palmas
  - Hospital de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital de la Princesa, Madrid
  - Complejo Hospitalario Santa Maria, Ourense
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Consorci Hospitalari del Parc Tauli, Sabadell
  - Hospital Universitario Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Nuestra Senora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universidad Virgen Del Rocio, Seville
  - Hospital Virgen Del La Salud, Toledo
  - Hospital General Universitario Valencia, Valencia
  - Complexo Hospitalario Xeral de Vigo, Vigo Pontevedra
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (6):
  - University Hospital of Linkoping, Linköping
  - University Hospital of Malmoe, Malmo
  - Sahlgrenska University Hospital - Molndal at Gothenburg University, Mölndal
  - Karolinska University Hospital - Huddinge, Stockholm
  - Umea Universitet, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (8):
  - Kantonspital Aarau, Aarau
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Spitaeler Chur AG, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital - St. Gallen, Sankt Gallen
  - UniversitaetsSpital Zuerich, Zurich
- Thailand (2):
  - Chulalongkorn University Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
- United Kingdom (13):
  - Bradford Hospitals NHS Trust, Bradford, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Saint Margaret's Hospital, Epping Essex, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital, Hull, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Imperial College of Medicine, London, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Airedale General Hospital, West Yorkshire, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England

REFERENCES:
- [Background] Jahanzeb M. Adjuvant trastuzumab therapy for HER2-positive breast cancer. Clin Breast Cancer. 2008 Aug;8(4):324-33. doi: 10.3816/CBC.2008.n.037. PMID 18757259
- [Background] Shiroiwa T, Fukuda T, Shimozuma K, Ohashi Y, Tsutani K. The model-based cost-effectiveness analysis of 1-year adjuvant trastuzumab treatment: based on 2-year follow-up HERA trial data. Breast Cancer Res Treat. 2008 Jun;109(3):559-66. doi: 10.1007/s10549-007-9679-4. Epub 2007 Jul 28. PMID 17661170
- [Result] Gianni L, Dafni U, Gelber RD, Azambuja E, Muehlbauer S, Goldhirsch A, Untch M, Smith I, Baselga J, Jackisch C, Cameron D, Mano M, Pedrini JL, Veronesi A, Mendiola C, Pluzanska A, Semiglazov V, Vrdoljak E, Eckart MJ, Shen Z, Skiadopoulos G, Procter M, Pritchard KI, Piccart-Gebhart MJ, Bell R; Herceptin Adjuvant (HERA) Trial Study Team. Treatment with trastuzumab for 1 year after adjuvant chemotherapy in patients with HER2-positive early breast cancer: a 4-year follow-up of a randomised controlled trial. Lancet Oncol. 2011 Mar;12(3):236-44. doi: 10.1016/S1470-2045(11)70033-X. Epub 2011 Feb 25. PMID 21354370
- [Result] Procter M, Suter TM, de Azambuja E, Dafni U, van Dooren V, Muehlbauer S, Climent MA, Rechberger E, Liu WT, Toi M, Coombes RC, Dodwell D, Pagani O, Madrid J, Hall M, Chen SC, Focan C, Muschol M, van Veldhuisen DJ, Piccart-Gebhart MJ. Longer-term assessment of trastuzumab-related cardiac adverse events in the Herceptin Adjuvant (HERA) trial. J Clin Oncol. 2010 Jul 20;28(21):3422-8. doi: 10.1200/JCO.2009.26.0463. Epub 2010 Jun 7. PMID 20530280
- [Result] Dowsett M, Procter M, McCaskill-Stevens W, de Azambuja E, Dafni U, Rueschoff J, Jordan B, Dolci S, Abramovitz M, Stoss O, Viale G, Gelber RD, Piccart-Gebhart M, Leyland-Jones B. Disease-free survival according to degree of HER2 amplification for patients treated with adjuvant chemotherapy with or without 1 year of trastuzumab: the HERA Trial. J Clin Oncol. 2009 Jun 20;27(18):2962-9. doi: 10.1200/JCO.2008.19.7939. Epub 2009 Apr 13. PMID 19364966
- [Result] Untch M, Gelber RD, Jackisch C, Procter M, Baselga J, Bell R, Cameron D, Bari M, Smith I, Leyland-Jones B, de Azambuja E, Wermuth P, Khasanov R, Feng-Yi F, Constantin C, Mayordomo JI, Su CH, Yu SY, Lluch A, Senkus-Konefka E, Price C, Haslbauer F, Suarez Sahui T, Srimuninnimit V, Colleoni M, Coates AS, Piccart-Gebhart MJ, Goldhirsch A; HERA Study Team. Estimating the magnitude of trastuzumab effects within patient subgroups in the HERA trial. Ann Oncol. 2008 Jun;19(6):1090-6. doi: 10.1093/annonc/mdn005. Epub 2008 Feb 21. PMID 18296421
- [Result] McCaskill-Stevens W, Procter M, Goodbrand J, et al.: Disease-free survival according to local immunohistochemistry for HER2 and central fluorescence in situ hydridization for patients treated with adjuvant chemotherapy with and without trastuzumab in the HERA (BIG 01-01) trial. [Abstract] Breast Cancer Res Treat 106 (1): A-71, S18, 2007.
- [Result] Smith I, Procter M, Gelber RD, Guillaume S, Feyereislova A, Dowsett M, Goldhirsch A, Untch M, Mariani G, Baselga J, Kaufmann M, Cameron D, Bell R, Bergh J, Coleman R, Wardley A, Harbeck N, Lopez RI, Mallmann P, Gelmon K, Wilcken N, Wist E, Sanchez Rovira P, Piccart-Gebhart MJ; HERA study team. 2-year follow-up of trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer: a randomised controlled trial. Lancet. 2007 Jan 6;369(9555):29-36. doi: 10.1016/S0140-6736(07)60028-2. PMID 17208639
- [Result] Suter TM, Procter M, van Veldhuisen DJ, Muscholl M, Bergh J, Carlomagno C, Perren T, Passalacqua R, Bighin C, Klijn JG, Ageev FT, Hitre E, Groetz J, Iwata H, Knap M, Gnant M, Muehlbauer S, Spence A, Gelber RD, Piccart-Gebhart MJ. Trastuzumab-associated cardiac adverse effects in the herceptin adjuvant trial. J Clin Oncol. 2007 Sep 1;25(25):3859-65. doi: 10.1200/JCO.2006.09.1611. Epub 2007 Jul 23. PMID 17646669
- [Result] Piccart-Gebhart MJ, Procter M, Leyland-Jones B, Goldhirsch A, Untch M, Smith I, Gianni L, Baselga J, Bell R, Jackisch C, Cameron D, Dowsett M, Barrios CH, Steger G, Huang CS, Andersson M, Inbar M, Lichinitser M, Lang I, Nitz U, Iwata H, Thomssen C, Lohrisch C, Suter TM, Ruschoff J, Suto T, Greatorex V, Ward C, Straehle C, McFadden E, Dolci MS, Gelber RD; Herceptin Adjuvant (HERA) Trial Study Team. Trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1659-72. doi: 10.1056/NEJMoa052306. PMID 16236737
- [Derived] Bae SJ, Moon S, Kook Y, Baek SH, Lee M, Kim JH, Ahn SG, Jeong J. Clinical relevance of clinical treatment score post-5 years (CTS5) in HR-positive, HER2-positive breast cancer. NPJ Breast Cancer. 2025 Apr 2;11(1):33. doi: 10.1038/s41523-025-00747-6. PMID 40175431
- [Derived] Yerushalmi R, Dong B, Chapman JW, Goss PE, Pollak MN, Burnell MJ, Levine MN, Bramwell VHC, Pritchard KI, Whelan TJ, Ingle JN, Shepherd LE, Parulekar WR, Han L, Ding K, Gelmon KA. Impact of baseline BMI and weight change in CCTG adjuvant breast cancer trials. Ann Oncol. 2017 Jul 1;28(7):1560-1568. doi: 10.1093/annonc/mdx152. PMID 28379421
- [Derived] Cameron D, Piccart-Gebhart MJ, Gelber RD, Procter M, Goldhirsch A, de Azambuja E, Castro G Jr, Untch M, Smith I, Gianni L, Baselga J, Al-Sakaff N, Lauer S, McFadden E, Leyland-Jones B, Bell R, Dowsett M, Jackisch C; Herceptin Adjuvant (HERA) Trial Study Team. 11 years' follow-up of trastuzumab after adjuvant chemotherapy in HER2-positive early breast cancer: final analysis of the HERceptin Adjuvant (HERA) trial. Lancet. 2017 Mar 25;389(10075):1195-1205. doi: 10.1016/S0140-6736(16)32616-2. Epub 2017 Feb 17. PMID 28215665
- [Derived] Loi S, Dafni U, Karlis D, Polydoropoulou V, Young BM, Willis S, Long B, de Azambuja E, Sotiriou C, Viale G, Ruschoff J, Piccart MJ, Dowsett M, Michiels S, Leyland-Jones B. Effects of Estrogen Receptor and Human Epidermal Growth Factor Receptor-2 Levels on the Efficacy of Trastuzumab: A Secondary Analysis of the HERA Trial. JAMA Oncol. 2016 Aug 1;2(8):1040-7. doi: 10.1001/jamaoncol.2016.0339. PMID 27100299
- [Derived] O'Sullivan CC, Bradbury I, Campbell C, Spielmann M, Perez EA, Joensuu H, Costantino JP, Delaloge S, Rastogi P, Zardavas D, Ballman KV, Holmes E, de Azambuja E, Piccart-Gebhart M, Zujewski JA, Gelber RD. Efficacy of Adjuvant Trastuzumab for Patients With Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer and Tumors </= 2 cm: A Meta-Analysis of the Randomized Trastuzumab Trials. J Clin Oncol. 2015 Aug 20;33(24):2600-8. doi: 10.1200/JCO.2015.60.8620. Epub 2015 Jun 22. PMID 26101239
- [Derived] de Azambuja E, Procter MJ, van Veldhuisen DJ, Agbor-Tarh D, Metzger-Filho O, Steinseifer J, Untch M, Smith IE, Gianni L, Baselga J, Jackisch C, Cameron DA, Bell R, Leyland-Jones B, Dowsett M, Gelber RD, Piccart-Gebhart MJ, Suter TM. Trastuzumab-associated cardiac events at 8 years of median follow-up in the Herceptin Adjuvant trial (BIG 1-01). J Clin Oncol. 2014 Jul 10;32(20):2159-65. doi: 10.1200/JCO.2013.53.9288. Epub 2014 Jun 9. PMID 24912899
- [Derived] Zabaglo L, Stoss O, Ruschoff J, Zielinski D, Salter J, Arfi M, Bradbury I, Dafni U, Piccart-Gebhart M, Procter M, Dowsett M; HERA Trial Study Team. HER2 staining intensity in HER2-positive disease: relationship with FISH amplification and clinical outcome in the HERA trial of adjuvant trastuzumab. Ann Oncol. 2013 Nov;24(11):2761-6. doi: 10.1093/annonc/mdt275. Epub 2013 Jul 25. PMID 23894039
- [Derived] Goldhirsch A, Gelber RD, Piccart-Gebhart MJ, de Azambuja E, Procter M, Suter TM, Jackisch C, Cameron D, Weber HA, Heinzmann D, Dal Lago L, McFadden E, Dowsett M, Untch M, Gianni L, Bell R, Kohne CH, Vindevoghel A, Andersson M, Brunt AM, Otero-Reyes D, Song S, Smith I, Leyland-Jones B, Baselga J; Herceptin Adjuvant (HERA) Trial Study Team. 2 years versus 1 year of adjuvant trastuzumab for HER2-positive breast cancer (HERA): an open-label, randomised controlled trial. Lancet. 2013 Sep 21;382(9897):1021-8. doi: 10.1016/S0140-6736(13)61094-6. Epub 2013 Jul 18. PMID 23871490
- [Derived] Metzger-Filho O, Procter M, de Azambuja E, Leyland-Jones B, Gelber RD, Dowsett M, Loi S, Saini KS, Cameron D, Untch M, Smith I, Gianni L, Baselga J, Jackisch C, Bell R, Sotiriou C, Viale G, Piccart-Gebhart M. Magnitude of trastuzumab benefit in patients with HER2-positive, invasive lobular breast carcinoma: results from the HERA trial. J Clin Oncol. 2013 Jun 1;31(16):1954-60. doi: 10.1200/JCO.2012.46.2440. Epub 2013 Apr 15. PMID 23589556

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the release of initial study results, participants in the Observation Arm without disease recurrence were given the opportunity to cross over to receive 1 or 2 years of adjuvant Herceptin. Efficacy analyses were still performed according to original randomization.
Groups:
- Observation Arm: Participants who completed definitive surgery and systemic adjuvant chemotherapy were observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant. No Herceptin was provided.
- Herceptin 1-Year Arm: Participants who completed definitive surgery and systemic adjuvant chemotherapy received a loading dose of Herceptin as 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion on Day 1, followed by a maintenance dose of 6 mg/kg via IV infusion 3 weeks later and thereafter every 3 weeks for 1 year or until disease recurrence, whichever occurred first. Participants were observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant.
- Herceptin 2-Year Arm: Participants who completed definitive surgery and systemic adjuvant chemotherapy received a loading dose of Herceptin as 8 mg/kg via IV infusion on Day 1, followed by a maintenance dose of 6 mg/kg via IV infusion 3 weeks later and thereafter every 3 weeks for 2 years or until disease recurrence, whichever occurred first. Participants were observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant.
Period: Overall Study
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Started | 1697 (Included all participants with available signed Informed Consent Form.) | 1702 (Included all participants with available signed Informed Consent Form.) | 1700 (Included all participants with available signed Informed Consent Form.)
Crossover to Adjuvant Herceptin | 888 | 0 (This milestone is not applicable to participants who were already randomized to Herceptin.) | 0 (This milestone is not applicable to participants who were already randomized to Herceptin.)
Completed | 834 | 994 | 974
Not Completed | 863 | 708 | 726
Not completed — Adverse Event/Intercurrent Illness | 2 | 2 | 7
Not completed — Death | 22 | 24 | 17
Not completed — Insufficient Therapeutic Response | 542 | 437 | 445
Not completed — Violation of Selection Criteria at Entry | 3 | 6 | 6
Not completed — Other Protocol Violation | 2 | 0 | 1
Not completed — Refused/Did Not Cooperate/Withdrew | 142 | 93 | 84
Not completed — Failure to Return | 57 | 62 | 61
Not completed — Other | 93 | 84 | 105

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) Population: All enrolled/randomized participants who had an available signed Informed Consent Form.
Groups:
- Herceptin 1-Year Arm: Participants who completed definitive surgery and systemic adjuvant chemotherapy received a loading dose of Herceptin as 8 mg/kg via IV infusion on Day 1, followed by a maintenance dose of 6 mg/kg via IV infusion 3 weeks later and thereafter every 3 weeks for 1 year or until disease recurrence, whichever occurred first. Participants were observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant.
- Total: Total of all reporting groups
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm | Total
Number analyzed (Participants) | 1697 | 1702 | 1700 | 5099
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.08) | 49.0 (10.06) | 49.2 (10.09) | 49.1 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1697 | 1702 | 1700 | 5099
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease-Free Survival (DFS) Events in Herceptin 1-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants with at least one DFS event was reported. The analysis of the Herceptin 1-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed by the Sponsor in 2006 following database cleaning. The analysis of the Herceptin 2-Year Arm against the Observation Arm was performed for an Independent Data Monitoring Committee (IDMC) in 2005 at a time the Sponsor was blinded. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: From Baseline until time of event (median of 1 year)
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm
Number analyzed (Participants) | 1693 | 1693
percentage of participants | 12.9 | 7.5
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.44 to 0.67] — HR for Herceptin 1-Year Arm versus Observation Arm

2. Primary Outcome: Percentage of Participants With DFS Events in Herceptin 2-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants with at least one DFS event was reported. The analysis of the Herceptin 2-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed for an IDMC in 2005 at a time the Sponsor was blinded. The analysis of the Herceptin 1-Year Arm against the Observation Arm was performed by the Sponsor in 2006 following database cleaning. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: From Baseline until time of event (median of 1 year)
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1693 | 1694
percentage of participants | 13.0 | 7.6
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.000, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.34 to 0.53] — HR for Herceptin 2-Year Arm versus Observation Arm

3. Primary Outcome: DFS Rate According to Kaplan-Meier Analysis in Herceptin 1-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants free of DFS events (i.e., the DFS rate) and corresponding 95 percent (%) confidence interval (CI) were estimated by Kaplan-Meier analysis based on available data at the time of the 1-year median follow-up analysis. The analysis of the Herceptin 1-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed by the Sponsor in 2006 following database cleaning. The analysis of the Herceptin 2-Year Arm against the Observation Arm was performed for an IDMC in 2005 at a time the Sponsor was blinded. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: Year 2
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm
Number analyzed (Participants) | 1693 | 1693
percentage of participants | 78.18 [75 to 81] | 85.80 [83 to 89]

4. Primary Outcome: DFS Rate According to Kaplan-Meier Analysis in Herceptin 2-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants free of DFS events (i.e., the DFS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 1-year median follow-up analysis. The analysis of the Herceptin 2-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed for an IDMC in 2005 at a time the Sponsor was blinded. The analysis of the Herceptin 1-Year Arm against the Observation Arm was performed by the Sponsor in 2006 following database cleaning. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: Year 2
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1693 | 1694
percentage of participants | 73.60 [70 to 77] | 87.50 [85 to 90]

5. Primary Outcome: Percentage of Participants With DFS Events Compared to Observation: 8-Year Median Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants with at least one DFS event was reported.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 33.6 | 27.7 | 27.8
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.67 to 0.86] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 3: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 4: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.67 to 0.85] — HR for Herceptin 2-Year Arm versus Observation Arm

6. Primary Outcome: DFS Rate at Year 3 According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants free of DFS events (i.e., the DFS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis.
Time Frame: Year 3
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 75.2 [73.1 to 77.3] | 81.3 [79.4 to 83.2] | 83.5 [81.7 to 85.3]

7. Primary Outcome: DFS Rate at Year 5 According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: as for outcome 6
Time Frame: Year 5
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 70.0 [67.8 to 72.3] | 75.9 [73.8 to 78.0] | 76.5 [74.4 to 78.5]

8. Primary Outcome: DFS Rate at Year 7 According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: as for outcome 6
Time Frame: Year 7
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 66.0 [63.6 to 68.3] | 72.4 [70.2 to 74.6] | 72.5 [70.4 to 74.7]

9. Primary Outcome: DFS Rate at Year 8 According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: as for outcome 6
Time Frame: Year 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 64.8 [62.4 to 67.2] | 71.2 [69.0 to 73.4] | 71.0 [68.7 to 73.2]

10. Primary Outcome: Percentage of Participants With DFS Events Compared to Observation: 10-Year Maximum Follow-Up
Description: as for outcome 5
Time Frame: From Baseline until time of event (maximum of 10 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 35.8 | 29.7 | 30.5
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.68 to 0.86] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.69 to 0.87] — HR for Herceptin 2-Year Arm versus Observation Arm

11. Primary Outcome: DFS Rate at Year 3 According to Kaplan-Meier Analysis Compared to Observation: 10-Year Maximum Follow-Up
Description: DFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer or second non-breast malignancy other than basal or squamous carcinoma of the skin and carcinoma in situ of the cervix, or death from any cause. The percentage of participants free of DFS events (i.e., the DFS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the final analysis with a 10-year maximum follow-up for DFS events.
Time Frame: Year 3
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 75.2 [73.1 to 77.3] | 81.3 [79.4 to 83.2] | 83.4 [81.6 to 85.2]

12. Primary Outcome: DFS Rate at Year 5 According to Kaplan-Meier Analysis Compared to Observation: 10-Year Maximum Follow-Up
Description: as for outcome 11
Time Frame: Year 5
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 70.0 [67.8 to 72.2] | 75.9 [73.8 to 78.0] | 76.4 [74.4 to 78.5]

13. Primary Outcome: DFS Rate at Year 7 According to Kaplan-Meier Analysis Compared to Observation: 10-Year Maximum Follow-Up
Description: as for outcome 11
Time Frame: Year 7
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 65.8 [63.5 to 68.2] | 72.4 [70.2 to 74.5] | 72.5 [70.3 to 74.7]

14. Primary Outcome: DFS Rate at Year 8 According to Kaplan-Meier Analysis Compared to Observation: 10-Year Maximum Follow-Up
Description: as for outcome 11
Time Frame: Year 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 64.7 [62.3 to 67.0] | 71.2 [69.0 to 73.4] | 70.7 [68.5 to 72.9]

15. Primary Outcome: DFS Rate at Year 9 According to Kaplan-Meier Analysis Compared to Observation: 10-Year Maximum Follow-Up
Description: as for outcome 11
Time Frame: Year 9
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 63.5 [61.2 to 65.9] | 70.3 [68.1 to 72.6] | 69.2 [67.0 to 71.5]

16. Primary Outcome: DFS Rate at Year 10 According to Kaplan-Meier Analysis Compared to Observation: 10-Year Maximum Follow-Up
Description: as for outcome 11
Time Frame: Year 10
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 62.5 [60.1 to 64.8] | 69.3 [67.0 to 71.5] | 68.5 [66.2 to 70.7]

17. Secondary Outcome: Percentage of Participants With DFS Events in 1-Year Versus 2-Year Herceptin: 10-Year Maximum Follow-Up
Description: as for outcome 5
Time Frame: From Baseline until time of event (maximum of 10 years)
Population: FAS Population 1-Year Herceptin Versus 2-Year Herceptin (1Y2Y): Participants without a DFS event and still under follow-up at the pre-defined landmark of 366 days after randomization, analyzed when intent-to-treat principle was applied for comparison of 1 year versus 2 years of Herceptin.
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 25.8 | 26.6
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.7962, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.89 to 1.17] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

18. Secondary Outcome: DFS Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 10-Year Maximum Follow-Up
Description: as for outcome 11
Time Frame: Years 3, 5, 7, 8, 9, 10
Population: FAS Population 1Y2Y
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 86.7 [85.0 to 88.4] | 89.0 [87.4 to 90.6]
  Year 5 | 81.0 [79.0 to 82.9] | 81.6 [79.6 to 83.5]
  Year 7 | 77.2 [75.1 to 79.3] | 77.4 [75.3 to 79.5]
  Year 8 | 75.9 [73.8 to 78.1] | 75.5 [73.3 to 77.7]
  Year 9 | 75.0 [72.8 to 77.2] | 73.9 [71.7 to 76.1]
  Year 10 | 73.9 [71.7 to 76.1] | 73.1 [70.8 to 75.3]

19. Secondary Outcome: Percentage of Participants With Overall Survival (OS) Events in Herceptin 1-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants who died was reported. The analysis of the Herceptin 1-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed by the Sponsor in 2006 following database cleaning. The analysis of the Herceptin 2-Year Arm against the Observation Arm was performed for an IDMC in 2005 at a time the Sponsor was blinded. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: From Baseline until time of event (median of 1 year)
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm
Number analyzed (Participants) | 1693 | 1693
percentage of participants | 2.4 | 1.8
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p = 0.2379, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.47 to 1.21] — HR for Herceptin 1-Year Arm versus Observation Arm

20. Secondary Outcome: Percentage of Participants With OS Events in Herceptin 2-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants who died was reported. The analysis of the Herceptin 2-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed for an IDMC in 2005 at a time the Sponsor was blinded. The analysis of the Herceptin 1-Year Arm against the Observation Arm was performed by the Sponsor in 2006 following database cleaning. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: From Baseline until time of event (median of 1 year)
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1693 | 1694
percentage of participants | 2.2 | 1.4
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.003, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.28 to 0.79] — HR for Herceptin 2-Year Arm versus Observation Arm

21. Secondary Outcome: OS Rate According to Kaplan-Meier Analysis in Herceptin 1-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants alive (i.e., the OS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 1-year median follow-up analysis. The analysis of the Herceptin 1-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed by the Sponsor in 2006 following database cleaning. The analysis of the Herceptin 2-Year Arm against the Observation Arm was performed for an IDMC in 2005 at a time the Sponsor was blinded. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: Year 2
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm
Number analyzed (Participants) | 1693 | 1693
percentage of participants | 94.98 [93 to 97] | 95.88 [94 to 98]

22. Secondary Outcome: OS Rate According to Kaplan-Meier Analysis in Herceptin 2-Year Arm Compared to Observation: 1-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants alive (i.e., the OS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 1-year median follow-up analysis. The analysis of the Herceptin 2-Year Arm against the Observation Arm after 1-year median follow-up, as reported below, was performed for an IDMC in 2005 at a time the Sponsor was blinded. The analysis of the Herceptin 1-Year Arm against the Observation Arm was performed by the Sponsor in 2006 following database cleaning. Therefore, these data are reported under a separate Outcome Measure.
Time Frame: Year 2
Population: FAS Population. The "Number of Participants Analyzed" reflects the number with data for the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1693 | 1694
percentage of participants | 94.39 [92 to 97] | 97.28 [96 to 98]

23. Secondary Outcome: Percentage of Participants With OS Events Compared to Observation: 8-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants who died was reported.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 20.6 | 16.3 | 16.1
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p = 0.0005, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.65 to 0.88] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 3: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.0001, Log Rank
Statistical Analysis 4: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.86] — HR for Herceptin 2-Year Arm versus Observation Arm

24. Secondary Outcome: OS Rate According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants alive (i.e., the OS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis.
Time Frame: Years 3, 5, 7, 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants
  Year 3 | 90.7 [89.3 to 92.1] | 92.7 [91.5 to 94.0] | 94.4 [93.3 to 95.6]
  Year 5 | 84.5 [82.8 to 86.3] | 86.9 [85.2 to 88.5] | 88.7 [87.2 to 90.3]
  Year 7 | 79.5 [77.5 to 81.5] | 83.9 [82.1 to 85.7] | 84.6 [82.9 to 86.4]
  Year 8 | 77.4 [75.2 to 79.5] | 82.7 [80.8 to 84.6] | 82.4 [80.4 to 84.3]

25. Secondary Outcome: Percentage of Participants With OS Events Compared to Observation: 11-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants who died was reported.
Time Frame: From Baseline until time of event (median of 11 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 23.9 | 18.8 | 18.4
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.64 to 0.86] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.62 to 0.83] — HR for Herceptin 2-Year Arm versus Observation Arm

26. Secondary Outcome: OS Rate According to Kaplan-Meier Analysis Compared to Observation: 11-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants alive (i.e., the OS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the final analysis with an 11-year median follow-up for OS events.
Time Frame: Years 3, 5, 7, 9, 10, 11, 12
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants
  Year 3 | 90.7 [89.3 to 92.1] | 92.7 [91.5 to 94.0] | 94.4 [93.3 to 95.6]
  Year 5 | 84.5 [82.8 to 86.3] | 86.9 [85.2 to 88.5] | 88.7 [87.2 to 90.3]
  Year 7 | 79.4 [77.4 to 81.4] | 83.8 [82.0 to 85.6] | 84.7 [82.9 to 86.4]
  Year 9 | 76.5 [74.4 to 78.6] | 81.9 [80.0 to 83.8] | 81.8 [80.0 to 83.7]
  Year 10 | 75.0 [72.9 to 77.2] | 80.7 [78.8 to 82.6] | 81.0 [79.0 to 82.9]
  Year 11 | 73.7 [71.5 to 76.0] | 80.0 [78.1 to 82.0] | 80.3 [78.3 to 82.3]
  Year 12 | 72.9 [70.4 to 75.3] | 79.4 [77.3 to 81.5] | 79.5 [77.4 to 81.7]

27. Secondary Outcome: Percentage of Participants With OS Events in 1-Year Versus 2-Year Herceptin: 11-Year Median Follow-Up
Description: OS events referred to death from any cause. The percentage of participants who died was reported.
Time Frame: From Baseline until time of event (median of 11 years)
Population: FAS Population 1Y2Y
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 14.7 | 14.9
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.9156, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.84 to 1.21] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

28. Secondary Outcome: OS Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 11-Year Median Follow-Up
Description: as for outcome 26
Time Frame: Years 3, 5, 7, 9, 10, 11, 12
Population: FAS Population 1Y2Y
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 96.5 [95.6 to 97.4] | 97.4 [96.6 to 98.2]
  Year 5 | 91.4 [90.0 to 92.8] | 92.6 [91.2 to 93.9]
  Year 7 | 88.6 [87.0 to 90.2] | 88.7 [87.1 to 90.3]
  Year 9 | 86.7 [85.0 to 88.5] | 85.9 [84.2 to 87.7]
  Year 10 | 85.4 [83.6 to 87.2] | 85.1 [83.3 to 86.9]
  Year 11 | 84.7 [82.9 to 86.6] | 84.4 [82.5 to 86.2]
  Year 12 | 84.1 [82.1 to 86.1] | 83.6 [81.5 to 85.6]

29. Secondary Outcome: Percentage of Participants With Recurrence-Free Survival (RFS) Events Compared to Observation: 8-Year Median Follow-Up
Description: RFS events included local, regional, or distant tumor recurrence. The percentage of participants with at least one RFS event was reported.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 29.8 | 23.4 | 22.6
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.64 to 0.83] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 3: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 4: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.61 to 0.79] — HR for Herceptin 2-Year Arm versus Observation Arm

30. Secondary Outcome: RFS Rate According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: RFS events included local, regional, or distant tumor recurrence. The percentage of participants free of RFS events (i.e., the RFS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis.
Time Frame: Years 3, 5, 7, 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants
  Year 3 | 76.4 [74.3 to 78.4] | 82.7 [80.9 to 84.6] | 86.0 [84.3 to 87.6]
  Year 5 | 71.9 [69.7 to 74.1] | 78.4 [76.4 to 80.4] | 79.9 [77.9 to 81.9]
  Year 7 | 69.0 [66.7 to 71.3] | 75.7 [73.6 to 77.8] | 76.7 [74.6 to 78.8]
  Year 8 | 68.4 [66.1 to 70.7] | 75.1 [72.9 to 77.2] | 75.8 [73.6 to 77.9]

31. Secondary Outcome: Percentage of Participants With RFS Events in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 29
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population 1Y2Y
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 19.7 | 18.8
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.4755, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.80 to 1.11] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

32. Secondary Outcome: RFS Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 30
Time Frame: Years 3, 5, 7, 8
Population: FAS Population 1Y2Y
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 87.7 [86.0 to 89.3] | 90.9 [89.4 to 92.3]
  Year 5 | 83.1 [81.2 to 85.0] | 84.5 [82.7 to 86.4]
  Year 7 | 80.2 [78.2 to 82.3] | 81.3 [79.3 to 83.2]
  Year 8 | 79.6 [77.5 to 81.6] | 80.3 [78.2 to 82.3]

33. Secondary Outcome: Percentage of Participants With Distant Disease-Free Survival (DDFS) Events Compared to Observation: 8-Year Median Follow-Up
Description: DDFS events included distant tumor recurrence, second primary cancer, or contralateral breast cancer. The percentage of participants with at least one DDFS event was reported.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 28.8 | 23.4 | 23.2
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.67 to 0.87] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 3: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 4: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.65 to 0.85] — HR for Herceptin 2-Year Arm versus Observation Arm

34. Secondary Outcome: DDFS Rate According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: DDFS events included distant tumor recurrence, second primary cancer, or contralateral breast cancer. The percentage of participants free of DDFS events (i.e., the DDFS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis.
Time Frame: Years 3, 5, 7, 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants
  Year 3 | 78.6 [76.6 to 80.6] | 84.4 [82.7 to 86.2] | 85.9 [84.2 to 87.6]
  Year 5 | 74.2 [72.1 to 76.4] | 79.6 [77.6 to 81.6] | 80.2 [78.2 to 82.1]
  Year 7 | 70.8 [68.6 to 73.1] | 76.7 [74.6 to 78.8] | 76.7 [74.6 to 78.8]
  Year 8 | 69.6 [67.3 to 71.9] | 75.5 [73.4 to 77.6] | 75.6 [73.4 to 77.7]

35. Secondary Outcome: Percentage of Participants With DDFS Events in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 33
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population 1Y2Y
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 19.5 | 19.5
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.9626, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.85 to 1.17] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

36. Secondary Outcome: DDFS Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 34
Time Frame: Years 3, 5, 7, 8
Population: FAS Population 1Y2Y
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 89.4 [87.9 to 91.0] | 90.8 [89.4 to 92.2]
  Year 5 | 84.5 [82.7 to 86.3] | 84.7 [82.9 to 86.5]
  Year 7 | 81.4 [79.5 to 83.4] | 81.1 [79.1 to 83.1]
  Year 8 | 80.1 [78.1 to 82.2] | 79.9 [77.8 to 81.9]

37. Secondary Outcome: Percentage of Participants With Tumor Recurrence (TR) Compared to Observation: 8-Year Median Follow-Up
Description: The percentage of participants with TR of the present breast cancer was reported. TR included local, regional, or distant tumor ignoring contralateral breast cancer and second non-breast malignancy.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 29.8 | 23.4 | 22.6
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.64 to 0.83] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 3: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 4: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.61 to 0.79] — HR for Herceptin 2-Year Arm versus Observation Arm

38. Secondary Outcome: TR-Free Rate According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: The percentage of participants without TR of the present breast cancer (i.e., the TR-free rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis. TR included local, regional, or distant tumor ignoring contralateral breast cancer and second non-breast malignancy.
Time Frame: Years 3, 5, 7, 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants
  Year 3 | 76.5 [74.4 to 78.5] | 82.8 [81.0 to 84.6] | 86.1 [84.4 to 87.7]
  Year 5 | 72.1 [69.9 to 74.3] | 78.6 [76.6 to 80.6] | 80.1 [78.2 to 82.1]
  Year 7 | 69.2 [67.0 to 71.5] | 75.9 [73.9 to 78.0] | 77.0 [75.0 to 79.1]
  Year 8 | 68.6 [66.4 to 70.9] | 75.3 [73.2 to 77.4] | 76.2 [74.1 to 78.3]

39. Secondary Outcome: Percentage of Participants With TR in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 37
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population 1Y2Y
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 19.7 | 18.8
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.4500, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.80 to 1.10] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

40. Secondary Outcome: TR-Free Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 38
Time Frame: Years 3, 5, 7, 8
Population: FAS Population 1Y2Y
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 87.7 [86.1 to 89.4] | 90.9 [89.5 to 92.4]
  Year 5 | 83.2 [81.3 to 85.1] | 84.7 [82.9 to 86.5]
  Year 7 | 80.4 [78.4 to 82.4] | 81.5 [79.6 to 83.5]
  Year 8 | 79.8 [77.7 to 81.8] | 80.6 [78.6 to 82.6]

41. Secondary Outcome: Percentage of Participants With Distant Tumor Recurrence (DTR) Compared to Observation: 8-Year Median Follow-Up
Description: The percentage of participants with DTR was reported. DTR included distant tumors ignoring local and regional recurrences, contralateral breast cancer, and second non-breast malignancy.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants | 25.3 | 19.4 | 18.8
Statistical Analysis 1: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Observation Arm vs Herceptin 1-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.62 to 0.83] — HR for Herceptin 1-Year Arm versus Observation Arm
Statistical Analysis 3: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 4: Comparison: Observation Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.59 to 0.79] — HR for Herceptin 2-Year Arm versus Observation Arm

42. Secondary Outcome: DTR-Free Rate According to Kaplan-Meier Analysis Compared to Observation: 8-Year Median Follow-Up
Description: The percentage of participants without DTR (i.e., the DTR-free rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis. DTR included distant tumors ignoring local and regional recurrences, contralateral breast cancer, and second non-breast malignancy.
Time Frame: Years 3, 5, 7, 8
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1697 | 1702 | 1700
percentage of participants
  Year 3 | 79.8 [77.8 to 81.7] | 85.9 [84.2 to 87.6] | 88.1 [86.5 to 89.6]
  Year 5 | 76.5 [74.4 to 78.5] | 82.1 [80.2 to 84.0] | 83.4 [81.5 to 85.2]
  Year 7 | 74.0 [71.8 to 76.1] | 80.1 [78.2 to 82.1] | 80.7 [78.8 to 82.6]
  Year 8 | 73.3 [71.1 to 75.5] | 79.5 [77.5 to 81.5] | 80.3 [78.3 to 82.2]

43. Secondary Outcome: Percentage of Participants With DTR in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 41
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population 1Y2Y
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 15.5 | 15.1
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.6823, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.80 to 1.15] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

44. Secondary Outcome: DTR-Free Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: as for outcome 42
Time Frame: Years 3, 5, 7, 8
Population: FAS Population 1Y2Y
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 90.5 [89.0 to 91.9] | 92.4 [91.1 to 93.8]
  Year 5 | 86.7 [85.0 to 88.4] | 87.5 [85.8 to 89.2]
  Year 7 | 84.6 [82.8 to 86.4] | 84.9 [83.1 to 86.7]
  Year 8 | 83.9 [82.1 to 85.8] | 84.4 [82.6 to 86.3]

45. Secondary Outcome: Percentage of Participants With Restricted Disease-Free Survival (RDFS) Events in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: RDFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer, or death from any cause. The percentage of participants with at least one RDFS event was reported.
Time Frame: From Baseline until time of event (median of 8 years)
Population: FAS Population 1Y2Y. In contrast to other study endpoints, RDFS compared to the Observation Arm was not a planned endpoint according to study protocol. Only RDFS in Herceptin 1-Year Arm versus Herceptin 2-Year Arm was a planned endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants | 22.2 | 21.9
Statistical Analysis 1: Comparison: Herceptin 1-Year Arm vs Herceptin 2-Year Arm; Test type: Superiority or Other; p = 0.7251, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.84 to 1.13] — HR for Herceptin 2-Year Arm versus Herceptin 1-Year Arm

46. Secondary Outcome: RDFS Rate According to Kaplan-Meier Analysis in 1-Year Versus 2-Year Herceptin: 8-Year Median Follow-Up
Description: RDFS events included loco-regional or distant recurrence of breast cancer, development of contralateral breast cancer, or death from any cause. The percentage of participants free of RDFS events (i.e., the RDFS rate) and corresponding 95% CI were estimated by Kaplan-Meier analysis based on available data at the time of the 8-year median follow-up analysis.
Time Frame: Years 3, 5, 7, 8
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1552 | 1553
percentage of participants
  Year 3 | 87.3 [85.6 to 89.0] | 89.9 [88.4 to 91.4]
  Year 5 | 81.9 [79.9 to 83.8] | 83.0 [81.1 to 84.9]
  Year 7 | 78.5 [76.4 to 80.6] | 78.9 [76.9 to 81.0]
  Year 8 | 77.2 [75.1 to 79.3] | 77.7 [75.5 to 79.8]

47. Secondary Outcome: Percentage of Participants With Primary Cardiac Endpoint Events Compared to Observation: 10-Year Maximum Follow-Up
Description: Primary cardiac endpoint events included the occurrence of any of the following between randomization and new therapy for recurrent disease: symptomatic New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF) confirmed by a cardiologist with a drop in left ventricular ejection fraction (LVEF) at least 10 percentage points from Baseline and to a value less than (<) 50%, and documentation of definite or probable cardiac death. Definite cardiac death included CHF, myocardial infarction, or primary arrhythmia. Probable cardiac death included unexpected sudden death within 24 hours of a cardiac event (syncope, cardiac arrest, chest pain, infarction, arrhythmia) without documented etiology. The percentage of participants with at least one primary cardiac endpoint event was reported. The 95% CI was calculated by the Pearson-Clopper method for a one-sample binomial.
Time Frame: From Baseline until time of event (maximum up to 10 years)
Population: Safety Population: All participants randomized/enrolled in the study according to actual treatment received. Hence, participants assigned to Herceptin who received no study treatment were analyzed in the Observation Arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1744 | 1682 | 1673
percentage of participants | 0.11 [0.01 to 0.41] | 1.07 [0.64 to 1.69] | 1.02 [0.59 to 1.62]

48. Secondary Outcome: Percentage of Participants With Secondary Cardiac Endpoint Events Compared to Observation: 10-Year Maximum Follow-Up
Description: Secondary cardiac endpoint events included NYHA Class I or II CHF with a drop in LVEF measured by multiple-gated acquisition or electrocardiogram, unless the subsequent assessment of LVEF indicated a return to levels that did not meet the definition of a significant LVEF drop. A significant LVEF drop was defined as an absolute reduction of at least 10 percentage points from Baseline and to a value <50%. The percentage of participants with at least one secondary cardiac endpoint event was reported, excluding those with both a primary and secondary cardiac endpoint event. The 95% CI was calculated by the Pearson-Clopper method for a one-sample binomial.
Time Frame: From Baseline until time of event (maximum up to 10 years)
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Number analyzed (Participants) | 1744 | 1682 | 1673
percentage of participants | 0.86 [0.48 to 1.41] | 4.40 [3.47 to 5.49] | 7.29 [6.09 to 8.64]

ADVERSE EVENTS:
Time Frame: From Baseline until end of treatment (maximum up to 2 years) with the exception of cardiac/cardiovascular events, second primary malignancies, pregnancies, and Herceptin-related adverse events (maximum up to 10 years)
Description: Analysis Population Description: Safety Population
Groups:
- Observation Arm: Participants who completed definitive surgery and systemic adjuvant chemotherapy were observed for efficacy and safety until 10 years from individual randomization and for survival until 10 years after enrollment of the last participant. No Herceptin was provided. After the release of initial study results, participants in the Observation Arm were allowed to cross over to receive adjuvant Herceptin prior to disease recurrence. As such, adverse events that occurred after crossover were not included in the safety analyses for this arm.
Arm/Group | Observation Arm | Herceptin 1-Year Arm | Herceptin 2-Year Arm
Serious Adverse Events (participants affected / at risk) | 143/1744 | 269/1682 | 344/1673
Other Adverse Events (participants affected / at risk) | 1076/1744 | 1389/1682 | 1440/1673
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation Arm (N=1744) | Herceptin 1-Year Arm (N=1682) | Herceptin 2-Year Arm (N=1673)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 2 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 19 | 24
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 4 | 4
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericarditis lupus (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Tooth hypoplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 1 | 3
Cataract (Eye disorders) | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 1 | 0
Breast complication associated with device (General disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 3 | 0
Chills (General disorders) | 0 | 4 | 1
Death (General disorders) | 0 | 1 | 0
Device breakage (General disorders) | 0 | 1 | 0
Device dislocation (General disorders) | 0 | 0 | 2
Device failure (General disorders) | 0 | 0 | 1
Device leakage (General disorders) | 0 | 0 | 1
Fat necrosis (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Granuloma (General disorders) | 1 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 2 | 0
Medical device pain (General disorders) | 0 | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 1
Multi-organ disorder (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 6
Sudden death (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 3 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 4
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 2 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 5 | 5
Device related infection (Infections and infestations) | 2 | 9 | 8
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 8 | 4
Extradural abscess (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Genital infection female (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Lymphangitis (Infections and infestations) | 0 | 1 | 1
Mastitis (Infections and infestations) | 2 | 2 | 2
Muscle abscess (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 4 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Spinal cord abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 2 | 3 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 4
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 27 | 36
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 8 | 8
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 3
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Retro-orbital neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 7
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebellar atrophy (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 3 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0
Paresis (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 7 | 1
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 11 | 22 | 29
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 2 | 1
Delusion (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 5
Major depression (Psychiatric disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 1 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 2 | 1
Breast dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Breast fibrosis (Reproductive system and breast disorders) | 3 | 5 | 1
Breast haematoma (Reproductive system and breast disorders) | 0 | 1 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Breast inflammation (Reproductive system and breast disorders) | 1 | 3 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 1
Breast necrosis (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 3 | 4 | 7
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 2
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 2 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2 | 1
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 2 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 2 | 4
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Mammoplasty (Surgical and medical procedures) | 1 | 0 | 0
Nerve block (Surgical and medical procedures) | 1 | 0 | 0
Aortic occlusion (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 4 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 1 | 2 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Microangiopathy (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 2
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observation Arm (N=1744) | Herceptin 1-Year Arm (N=1682) | Herceptin 2-Year Arm (N=1673)
Cardiac failure congestive (Cardiac disorders) | 18 | 78 | 127
Palpitations (Cardiac disorders) | 20 | 72 | 84
Diarrhoea (Gastrointestinal disorders) | 22 | 155 | 180
Nausea (Gastrointestinal disorders) | 37 | 134 | 157
Vomiting (Gastrointestinal disorders) | 15 | 77 | 99
Asthenia (General disorders) | 42 | 102 | 119
Chest pain (General disorders) | 37 | 63 | 84
Chills (General disorders) | 1 | 99 | 128
Fatigue (General disorders) | 83 | 198 | 246
Oedema peripheral (General disorders) | 49 | 82 | 101
Pyrexia (General disorders) | 12 | 116 | 145
Influenza (Infections and infestations) | 17 | 95 | 142
Nasopharyngitis (Infections and infestations) | 65 | 187 | 269
Upper respiratory tract infection (Infections and infestations) | 31 | 53 | 84
Arthralgia (Musculoskeletal and connective tissue disorders) | 152 | 225 | 246
Back pain (Musculoskeletal and connective tissue disorders) | 106 | 146 | 137
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 69 | 91
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 64 | 70 | 92
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 88 | 104
Pain in extremity (Musculoskeletal and connective tissue disorders) | 74 | 97 | 107
Dizziness (Nervous system disorders) | 40 | 82 | 89
Headache (Nervous system disorders) | 72 | 201 | 250
Depression (Psychiatric disorders) | 59 | 88 | 80
Insomnia (Psychiatric disorders) | 49 | 96 | 75
Cough (Respiratory, thoracic and mediastinal disorders) | 62 | 116 | 147
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 83 | 116
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 52 | 83
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 53 | 98
Rash (Skin and subcutaneous tissue disorders) | 25 | 99 | 135
Hot flush (Vascular disorders) | 130 | 166 | 159
Hypertension (Vascular disorders) | 61 | 104 | 128
Lymphoedema (Vascular disorders) | 70 | 81 | 92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.